CLINICAL TRIAL: NCT04144725
Title: Ruling Out Coronary Artery Disease and Myocardial Injury by BiOmarkers: Light'n Easy
Brief Title: Ruling Out Coronary Artery Disease and Myocardial Injury by Biomarkers
Acronym: ROCAMBOLE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Torbjorn Omland, Professor, University Hospital, Akershus
Other Study IDs: 2017/1874
Record Dates: First submitted 2019-05-03; First posted 2019-10-30 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be obtained by venipuncture by dedicated study personnel in relation to the routine pre-procedural clinical examination conducted the same day or the day before the CCTA. The samples will be left at room temperature to coagulate and subsequently centrifuged at ~1500g for 15 minutes, and the supernatant will be transferred to acid-handled plastic tubes and analyzed directly or stored at -80℃.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected coronary artery disease: Patients hospitalized for suspected acute coronary syndrome who are referred to CCTA or patients referred to CCTA from outpatient clinics for evaluation of stable coronary artery disease.

SUMMARY:
A considerable proportion of patients with clinically suspected coronary artery disease (CAD) do not have angiographic signs of luminal narrowing caused by coronary atherosclerosis. In patients with suspected CAD, we will assess the ability of cardiovascular biomarkers to identify patients with (a) angiographically normal epicardial coronary vessels (b) absence of significant epicardial coronary stenosis, as assessed by coronary computed tomography angiography (CCTA). Patients will be stratified according to the presence or absence of dynamic changes of high sensitivity cardiac troponin T levels above the 99th percentile.

DETAILED DESCRIPTION:
This is an observational study of patients with suspected coronary artery disease referred to coronary computed tomography angiography (CCTA). The plan is to include 1000 patients prior to CCTA at two centers.

Blood samples for biomarker measurement will be obtained prior to the procedures. The diagnostic results of the imaging tests will be compared to the levels of circulating troponins. Patient will be followed for a minimum of 12 months and the incidence of cardiovascular death, all-cause mortality, acute coronary syndromes, revascularization, heart failure, stroke and cardiac arrhythmias requiring rehospitalization. Symptoms of angina pectoris according to the Canadian Cardiovascular Society grading of angina pectoris and symptoms of chronic heart failure according to the New York Heart Association classification of chronic heart failure will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Consenting patient over the age of 18 referred to CCTA for suspected coronary artery disease

Exclusion Criteria:

* Inability to provide informed consent.
* Short life expectancy (<12 months) due to non-cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational study of patients with suspected coronary artery disease referred to either emergent or out-patient coronary computed tomography angiography (CCTA)
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-10-23 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
The presence of obstructive coronary artery stenosis defined as diameter > 50% on CCTA | 0 days (Cross-sectional)
  Diagnostic end-point

SECONDARY OUTCOMES:
The presence of non-obstructive coronary artery stenosis defined as diameter stenosis 30-50% on CCTA | 0 days (Cross-sectional)
  Diagnostic end-point
Composite of cardiovascular death and hospitalization for heart failure or acute coronary syndrome | Follow-up until 2030
  Prognostic end-point
Incidence of cardiovascular death, hospitalization for myocardial infarction, unstable angina, revascularization, stroke, heart failure and cardiac arrhythmias. | Follow-up until 2030
  Prognostic-end-point

CONTACTS AND LOCATIONS:
Overall Officials: Torbjørn Omland, MD, PhD, Principal Investigator — University Hospital, Akershus
Locations (1):
- Akershus University Hospital, Lørenskog, Norway

IPD SHARING:
Plan to Share IPD: No